CLINICAL TRIAL: NCT04147351
Title: A Phase II Study of Atezolizumab in Combination With Bevacizumab, Carboplatin or Cisplatin, and Pemetrexed for EGFR-mutant Metastatic Non-small Cell Lung Cancer Patients After Failure of EGFR Tyrosine Kinase Inhibitors.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201908090MIFA
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: NSCLC Stage IIIB~IV
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab+bevacizumab+pemetrexed+carboplatin or cisplatin (Experimental)
  Interventions: Drug: Atezolizumab Injection; bevacizumab Injection

INTERVENTIONS:
Drug: Atezolizumab Injection; bevacizumab Injection — a PD-L1 inhibitor; anti-angiogenesis

SUMMARY:
using Atezolizumab, a PD-L1 inhibitor, in combination with bevacizumab, platinum and pemetrexed to treat patients with EGFR mutated, advanced non-small cell lung cancer (NSCLC) after failure of EGFR tyrosine kinase inhibitors.

DETAILED DESCRIPTION:
Patients diagnosed with (i) stage IIIB~IV non-small cell lung cancer, (ii) tumor harbors activating mutation at EGFR, (iii) radiological confirmation of progressive disease with one or more lines of EGFR tyrosine kinase inhibitors but have not yet been exposed to palliative chemotherapy, will be eligible for screening procedure. The lung cancer stage will be determined according to the 8th edition of the International Association for the Study of Lung Cancer (IASLC) Tumor, Node, Metastasis (TNM) staging system for lung cancer.

In addition to screening of baseline bone marrow function, organ functions, and CT assessment of measurable target lesion(s), patients after TKI treatment failure must receive tumor EGFR genotyping by testing tumor DNA in re-biopsied tumor samples. Testing report from local laboratories will be accepted.

Enrollment of patients into the study will depend on EGFR testing results in re-biopsied tumor samples.

Duration induction phase, four cycles of atezolizumab 1200 mg will be administered over 60 min (1st cycle) and 30 min (2nd cycle onwards); bevacizumab 7.5mg/kg over 90 min in 1st cycle, 60 min in 2nd cycle and 30 min in 3rd cycle onward; pemetrexed 500 mg/m2 over 10 min; and cisplatin 75mg/m2 or carboplatin (CCr < 60) area under curve 5 mg/mL per min over 15-60 min intravenously every 3 weeks in the order listed.

Following the induction phase, patients will continue atezolizumab, bevacizumab and pemetrexed as maintenance therapy. Patients will continue treatment with bevacizumab and pemetrexed until progressive disease, unacceptable toxicity, or death. Patients may continue treatment with atezolizumab beyond radiographic progression by RECIST v1.1, provided they are experiencing clinical benefit as assessed by investigator (i.e., in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data, biopsy results [if available], and clinical status.

Atezolizumab and bevacizumab dose reduction will not be allowed. Modification of carboplatin or cisplatin, and pemetrexed doses will be done according to the local guidelines of National Taiwan University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB~IV NSCLC with known EGFR activating mutation not amenable to curative surgery or radiotherapy. EGFR activating mutations include exon19 deletion, L858R, G719X, L861Q, or S768I.
* Radiological documentation of disease progression following one or more lines of EGFR TKI treatment but have not received palliative chemotherapy.
* Patients must receive tumor EGFR genotyping in re-biopsied FFPE tumor samples.
* At least 20 years of age.
* World Health Organisation (WHO) performance status 0-2 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computed tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
* Normal bone marrow and organ function as defined below:

  * Marrow: Hemoglobin ≥10gm/dL, absolute granulocyte count (AGC) ≥1500/mm3 platelets ≥100,000/mm3, absolute lymphocyte count ≥1000/mm3.
  * Hepatic: Serum/plasma total bilirubin ≤1.5 x upper limit of normal (ULN) with the exception of <2.9 mg/dL for patients with Gilbert's disease, ALT (SGPT) and AST (SGOT) ≤2.5 x ULN.
  * Renal: Serum/plasma creatinine (sCr) ≤1.5 x upper limit of normal, or creatinine clearance (Ccr) ≥45 mL/min.
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of atezolizumab and/or 6 months after the last dose of bevacizumab. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.

Exclusion Criteria:

* Previous exposure to platinum-based palliative chemotherapy. The treatment-free interval of neoadjuvant or adjuvant platinum-based chemotherapy should be more than 6 months before study enrollment is allowed
* Previous exposure to VEGF inhibitor for anti-cancer treatment
* Prior treatment with any other anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2) agent or an antibody targeting other immuno-regulatory receptors or mechanisms
* Patients carries EGFR genotype T790M or exon20 insertion should be excluded.
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of administration of atezolizumab.
* Expected to require any other form of antineoplastic therapy while on study
* Patients with untreated symptomatic brain metastases. Patients with treated brain metastases will be allowed if brain imaging obtained greater than 7 days from trial enrollment reveals stable disease. Patients with small (< 3mm) asymptomatic brain metastasis are allowed to enroll. Patients on steroids doses higher than 10 mg of prednisone (or its equivalent) are excluded
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to study enrollment.
* Leptomeningeal disease
* Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for locoregional therapy, if appropriate, prior to study enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX®) are allowed.
* Malignancies other than NSCLC within 5 years prior to study enrollment, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* On chronic systemic steroid therapy or on any other form of immunosuppressive medication
* Has received a live-virus vaccination within 30 days of planned treatment start
* Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, or abdominal carcinomatosis (known risks factors for bowel perforation)
* Severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* Active autoimmune disease that has required systemic treatment in the past 2 years (replacement therapies for hormone deficiencies are allowed) (see Appendix V)
* Systemic cytotoxic chemotherapy, antineoplastic biologic therapy, or major surgery within 3 weeks of the first dose of study medication
* Active infection requiring therapy
* History of Human Immunodeficiency Virus (HIV) unless recent serology test is negative.
* Hepatitis B carrier: Patients with HBV infection were required to be receiving effective antiviral therapy and have a viral load less than 100 IU/mL at screening
* Active Hepatitis C
* Interstitial lung disease or pneumonitis requiring oral or IV glucocorticoids
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable.
* History of hemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 9 MONTHS
  The percentage of patients with radiologically complete or partial response as determined by the investigator according to RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | about 9 months
  PFS is measured from the date of study enrollment to radiographically documented progression according to RECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan